CLINICAL TRIAL: NCT01462695
Title: A Phase II Study of Sunitinib (NSC# 736511) in Recurrent, Refractory or Progressive High Grade Glioma and Ependymoma Tumors in Pediatric and Young Adult Patients
Brief Title: Sunitinib Malate in Treating Younger Patients With Recurrent, Refractory, or Progressive Malignant Glioma or Ependymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03536; NCI-2011-03536 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000712861; COG-ACNS1021; ACNS1021 (Other: Children's Oncology Group); ACNS1021 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-06

CONDITIONS: Childhood Cerebellar Anaplastic Astrocytoma; Childhood Cerebral Anaplastic Astrocytoma; Childhood Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Mixed Glioma; Childhood Oligodendroglioma; Childhood Supratentorial Ependymoma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Familial ependymoma | interventions — Sunitinib

ARMS (1):
- Treatment (sunitinib) (Experimental): Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sunitinib Malate

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial studies how well sunitinib malate works in treating younger patients with recurrent, refractory, or progressive malignant glioma or ependymoma. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the objective response rate (partial response [PR] or complete response [CR] ≥ 8 weeks) to sunitinib in 2 strata (recurrent/progressive/refractory high-grade glioma vs ependymoma) of recurrent or progressive brain tumors in pediatric and young adult patients.

SECONDARY OBJECTIVES:

I. To explore and report descriptively the safety and tolerability of sunitinib in pediatric and young adult brain tumor patients who have not received prior anthracycline or radiotherapy involving the heart.

II. To describe the pharmacokinetic profile of pediatric and young adult patients taking sunitinib malate.

III. To describe the cumulative toxicities of sunitinib when administered over multiple courses to pediatric and young adult patients.

IV. To estimate progression-free survival (PFS) distributions for these cohorts of patients.

V. To evaluate changes in phosphorylation of PDGFR-α and -β, MEK/ERK, S6 kinase, and AKT in peripheral blood mononuclear cells and explore possible associations between these changes and outcome measures.

VI. To evaluate plasma levels of soluble isoforms of VEGFR-1 and -2 prior to initiation of therapy and at points during therapy as an exploration of possible biomarkers of clinical response.

VII. To evaluate and report descriptively the expression and ratio of VEGF isoforms in tumor tissue, as available.

VIII. To evaluate and report descriptively the genotype, expression, and possible amplification of KIT and PDGFR-α and -β in tumor tissue, as available.

OUTLINE: This is a multicenter study.

Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood sample collection at baseline and during courses 1 and 2 for pharmacokinetic and pharmacodynamic studies. Tissue samples from diagnosis and surgical resection may be also collected.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with ependymoma or high-grade glioma (World Health Organization [WHO] grade III/IV):

  * Stratum A: recurrent/progressive/refractory malignant glioma (i.e., anaplastic astrocytoma, glioblastoma multiforme [including giant cell and gliosarcoma types], anaplastic oligodendroglioma, anaplastic oligoastrocytoma, or anaplastic ganglioglioma) within the brain with or without spinal cord disease
  * Stratum B: recurrent/progressive/refractory ependymoma (including ependymoma variants) within the brain with or without spinal cord disease
  * Patients with diffuse intrinsic pontine glioma are not eligible
* A histological diagnosis from either the initial presentation or at the time of recurrence is required
* Patients must have radiographically documented measurable disease in the brain, defined as at least one lesion that can be accurately measured in at least 2 planes
* To document the degree of residual tumor, the following must be obtained:

  * All patients must have a brain MRI with and without gadolinium and a spine magnetic resonance imaging (MRI), if clinically indicated,with and without gadolinium, performed within 2 weeks prior to study enrollment
  * Patients with evidence of new central nervous system (CNS) hemorrhage of more than punctate size and/or more than 3 foci of punctate hemorrhage on baseline MRI obtained within 14 days prior to study enrollment are not eligible
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2 (use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age)

  * Neurological deficits in patients must have been relatively stable for a minimum of 1 week prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Peripheral absolute neutrophil count (ANC) ≥ 1,000/μL
* Platelet count ≥ 75,000/μL (transfusion independent, defined as not receiving platelet transfusions within the 7-day period prior to enrollment)
* Hemoglobin ≥ 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT/AST) and serum glutamic pyruvic transaminase (SGPT/ALT) ≤ 2.5 times ULN
* Shortening fraction of ≥ 27% by echocardiogram OR ejection fraction of ≥ 50% by radionuclide angiogram
* Corrected QT interval < 450 msec (males) or < 470 msec (females)
* Prothrombin time (PT) / international normalized ratio (INR) ≤ 1.5 times ULN
* Partial thromboplastin time (PTT) ≤ 1.5 times ULN
* Patients must not have a history of cardiac disease including, but not limited to:

  * Uncontrolled hypertension within 12 months prior to enrollment; uncontrolled hypertension is defined as follows:

    * Patients aged ≤ 17 years: greater than 95th percentile systolic and diastolic blood pressure based on age and height which is not controlled by one anti-hypertensive medication
    * Patients aged > 17 years: systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg which is not controlled by one anti-hypertensive medication
  * Ongoing cardiac dysrhythmias ≥ grade 2 or atrial fibrillation of any grade
  * Unstable angina, symptomatic congestive heart failure, or myocardial infarction
* Patients with a seizure disorder may be enrolled if on non-enzyme-inducing anticonvulsants and well controlled

  * Commonly used non-enzyme-inducing anticonvulsants include: gabapentin, lamotrigine, levetiracetam, tiagabine, topiramate, valproic acid, and zonisamide
* Patients must not have had a cerebrovascular accident or transient is chemic attack within 12 months prior to enrollment
* Patients must not have had a pulmonary embolism or other significant thromboembolic event within 12 months prior to enrollment
* Patients must not have had grade ≥ 3 hemorrhage within 4 weeks prior to enrollment
* Patients must not have had any of the following diagnoses within 6 months prior to enrollment: peptic ulcer disease, inflammatory bowel disease, or diverticulitis
* Patients with a diagnosis of abdomen fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to enrollment are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients with hypothyroidism that has not been well-controlled by medications for at least 2 weeks prior to study entry are not eligible
* Patients who have a personal history of genetic and/or congenital cardiac abnormalities are not eligible
* Patients who have a history of allergic reactions to compounds of similar chemical or biological composition to sunitinib are not eligible
* Patients who have any other condition that could result in an inability to swallow capsules/sprinkles or absorb oral sunitinib administered through a gastric tube are not eligible
* Patients with body surface area < 0.55 m^2 or > 2.18 m^2 are not eligible
* Female patients who are pregnant are not eligible
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained within the past 4 weeks
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation
* No concurrent use of nonsteroidal anti-inflammatory drugs (NSAIDs), clopidogrel, warfarin, heparin, low molecular weight heparin, dipyridamole, or aspirin therapy > 81 mg/day
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy (RT) prior to entering this study
* Must not have received myelosuppressive chemotherapy within 3 weeks of entry onto this study (6 weeks if prior nitrosourea)
* At least 7 days since the completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
* At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
* At least 24 weeks must have elapsed if prior full-field RT

  * ≥ 2 weeks must have elapsed if prior local palliative RT (small port) or limited-field RT
  * ≥ 3 months must have elapsed since prior stem cell transplant (SCT) or rescue with total-body irradiation (TBI)

    * No evidence of active graft-vs-host disease
* Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 7 days prior to enrollment
* Patients must not have received potent cytochrome P450-3A4 (CY3A4) inhibitors and/or inducers within 7 days prior to study enrollment and potent inducers within 12 days prior to study enrollment and during study
* At least 7 days must have elapsed since the completion of therapy with a hematopoietic growth factor
* Patients who have previously received sunitinib or who have received other VEGF-, PDGFR-, or KIT-targeted therapy are not eligible

  * Patients who received bevacizumab as part of their prior therapy may enroll on study
* Patients must not have received more than 2 prior chemotherapy and/or RT regimens; for example, 1 initial treatment course of chemotherapy and/or RT (counts as 1 treatment course) and at relapse may have received 1 treatment course of chemotherapy and/or RT (counts as 1 treatment course)
* Patients who received prior therapy with known risk for cardiovascular complications (e.g., anthracycline therapy or prior RT that included the heart and/or craniospinal radiation) are not eligible
* Patients receiving ongoing treatment with therapeutic doses (i.e., therapeutic INR levels) of coumarin derivatives or oral anti-vitamin K agents are not eligible
* Patients receiving antiretroviral therapy for human immunodeficiency virus (HIV) disease are not eligible
* Patients who are started on protocol therapy on a phase II study prior to study enrollment are considered ineligible
* No other concurrent chemotherapy, investigational agents, or immunomodulating agents
* No concurrent RT

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Wetmore, Principal Investigator — Children's Oncology Group
Locations (96):
- United States (86):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Issac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (5):
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

REFERENCES:
- [Derived] Wang E, DuBois SG, Wetmore C, Verschuur AC, Khosravan R. Population Pharmacokinetics of Sunitinib and its Active Metabolite SU012662 in Pediatric Patients with Gastrointestinal Stromal Tumors or Other Solid Tumors. Eur J Drug Metab Pharmacokinet. 2021 May;46(3):343-352. doi: 10.1007/s13318-021-00671-7. Epub 2021 Apr 14. PMID 33852135
- [Derived] Wang E, DuBois SG, Wetmore C, Khosravan R. Population pharmacokinetics-pharmacodynamics of sunitinib in pediatric patients with solid tumors. Cancer Chemother Pharmacol. 2020 Aug;86(2):181-192. doi: 10.1007/s00280-020-04106-z. Epub 2020 Jul 4. PMID 32623479
- [Derived] Wetmore C, Daryani VM, Billups CA, Boyett JM, Leary S, Tanos R, Goldsmith KC, Stewart CF, Blaney SM, Gajjar A. Phase II evaluation of sunitinib in the treatment of recurrent or refractory high-grade glioma or ependymoma in children: a children's Oncology Group Study ACNS1021. Cancer Med. 2016 Jul;5(7):1416-24. doi: 10.1002/cam4.713. Epub 2016 Apr 25. PMID 27109549

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum A: Recurrent High Grade Glioma; Stratum B: Recurrent Ependymoma: Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  sunitinib malate: Given PO
  diagnostic laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Stratum A: Recurrent High Grade Glioma | Stratum B: Recurrent Ependymoma
Started | 17 | 13
Completed | 0 | 0
Not Completed | 17 | 13
Not completed — Adverse Event | 1 | 1
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 6 | 12
Not completed — Physician Decision | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Inevaluable (did not receive study drug) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum A: Recurrent High Grade Glioma | Stratum B: Recurrent Ependymoma | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Median (Full Range); unit: years] | 14.2 [4.7 to 19.9] | 12.0 [3.0 to 16.9] | 13.4 [3.0 to 19.9]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 13 | 29
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 13 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 27
  Canada | 1 | 0 | 1
  Australia | 0 | 1 | 1
  Saudi Arabia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Sustained Objective Response Rate
Description: Sustained objective response was defined as a PR (Partial Response: ≥ 50% decrease in the sum of the products of the 2 perpendicular diameters of all target lesions (up to 5), taking as reference the initial baseline measurements) or CR (Complete Response: disappearance of all target lesions) lasting at least 8 weeks.
Time Frame: Up to 5 years
Population: One patient in Stratum A was excluded because the patient did not receive study drug and therefore was not evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Stratum A: Recurrent High Grade Glioma | Stratum B: Recurrent Ependymoma
Number analyzed (Participants) | 16 | 13
percentage of patients | 0 [0 to 19.8] | 0 [0 to 22.5]

ADVERSE EVENTS:
Description: One stratum A patient did not receive any study drug and was excluded from the summary of adverse events. SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs) or grade 5 adverse events resulting in death. The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Groups:
- Stratum B: Recurrent Ependymoma: Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Stratum A: Recurrent High Grade Glioma | Stratum B: Recurrent Ependymoma
Serious Adverse Events (participants affected / at risk) | 14/16 | 9/13
Other Adverse Events (participants affected / at risk) | 8/16 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A: Recurrent High Grade Glioma (N=16) | Stratum B: Recurrent Ependymoma (N=13)
Death NOS (General disorders) | 6 | 4
Gait disturbance (General disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5
Dysarthria (Nervous system disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 2 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A: Recurrent High Grade Glioma (N=16) | Stratum B: Recurrent Ependymoma (N=13)
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 5
Serum amylase increased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less